CLINICAL TRIAL: NCT06116370
Title: Two-Year Follow-Up Comparing Rezūm Therapy Versus Bipolar Transurethral Resection of the Prostate for Treating Benign Prostatic Hyperplasia. A Prospective Randomized Study.
Brief Title: The Clinical Efficacy of Rezūm Therapy Versus Bipolar Trans-urethral Resection of the Prostate for Treatment Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: surgical treatments of BPH
Record Dates: First submitted 2023-10-20; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-09

CONDITIONS: Prostatic Hyperplasia
Keywords: Rezum; LUTS; B-TURP
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPH patients treated with Rezum procedure (Active Comparator): Patients aged 50-80 years with prostate volumes of 50-120 ml, sexually active, and have severe LUTS treated with Rezum procedure
  Interventions: Procedure: Rezum procedure
- BPH patients treated with B-TURP procedure (Active Comparator): Patients aged 50-80 years with prostate volumes of 50-120 ml, sexually active, and have severe LUTS treated with Rezum procedure
  Interventions: Procedure: B-TURP procedure

INTERVENTIONS:
Procedure: Rezum procedure — In Rezūm procedure, the Rezūm System (NxThera Inc., Maple Grove, MN, USA) consists of a radiofrequency (RF) power supply generator and single-use transurethral delivery device. Starting 1 cm distal to the bladder neck, injection was done at 3 and 9 o'clock sites. The needle was inserted for 9 s duration, retracted, and then delivered to another treatment site in 1 cm distance distal to the previous one.
  Arms: BPH patients treated with Rezum procedure
Procedure: B-TURP procedure — In B-TURP, Olympus SurgMaster™ UES-40 bipolar generator (Olympus Europe, Hamburg, Germany) was used. Current's settings used were cut/coag 200/120. Using continuous flow 26Fr resectoscope first resection of the median lobe from the level of the bladder neck to the apex of the prostate was done followed by resection of the lateral lobes. Using Ellic evacuator, Prostatic chips were extracted from the field. A 22 fr three-way silicon Foley catheter was placed with traction applied and the balloon inflated by normal saline of 30-80 cc according to the size of the prostate.
  Arms: BPH patients treated with B-TURP procedure

SUMMARY:
We aimed to compare the efficacy and safety of Rezūm therapy and bipolar transurethral resection of prostate (B-TURP) for the management of benign prostatic hyperplasia (BPH) of 50-120gm size.

DETAILED DESCRIPTION:
For decades, Transurethral resection of the prostate (TURP) was the gold standard surgical intervention for small and moderate prostates, however it has high morbidity and prolonged hospital stay. In contrast to monopolar TURP (M-TURP), where prolonged resection carries the risk of transurethral resection (TUR) syndrome, bipolar transurethral resection of prostate (B-TURP), especially in large prostates was a promising procedure for urologists, but unfortunately, the morbidity rate of B-TURP remains high [4]. Therefore, newer minimally invasive procedures have been introduced to provide alternative surgical options to TURP.

Rezūm is a radiofrequency made water vapour thermal treatment. It has recently been added to the international guidelines as a choice for medical treatment resistant lower urinary tract symptoms (LUTS). The AUA and Canadian Urological Association (CUA) guidelines now add water vapour therapy as a treatment option for BPH patients with small prostate size <80 gm and for those wishing to maintain antegrade ejaculation. While they still offer no clear recommendation to Rezūm use for those with large prostates. Early studies on this topic have found out promising results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-80 years
* prostate volumes of 50-120 ml
* sexually active
* severe LUTS
* [Q max] of <10 ml/s
* [IPSS] of >20)
* failed medical treatment with alpha blockers

Exclusion Criteria:

* prostate cancer
* Neurogenic bladder
* urethral stricture
* urinary bladder stone
* previous prostatic surgery.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — disease specific to men
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Measurement of The International Prostate Symptom score (IPSS) in both groups | for each case in both groups the investigator assess IPSS at 6, 12, and 24 months after procedures through study completion, an average of 2 years
  After 6, 12, and 24 months of operation, the questioner is performed. Minimum :0 / Maximum : 35 Total score: 0-7 Mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic
Measurement of The Quality of Life (QoL) in both groups | for each case in both groups the investigator assess QoLat 6, 12, and 24 months after procedures through study completion, an average of 2 years
  After 6, 12, and 24 months of operation, the questioner is performed. Minimum :0 means delighted / Maximum : 5 means unhappy
Measurement of The Maximum Urinary flow rate (Qmax) in both groups | for each case in both groups the investigator assess Qmax at 6, 12, and 24 months after procedures through study completion, an average of 2 years
  After 6, 12, and 24 months of operation, the procedure is performed. Qmax is measured by (ml/sec) Normal values are described as a Qmax above 15 ml/sec and below 10 ml/sec is considered abnormal
Concentration of The Prostatic specific antigen (PSA) in both groups | for each case in both groups the investigator measures PSA at 6, 12, and 24 months after procedures through study completion, an average of 2 years
  After 6, 12, and 24 months of operation, the procedure is performed. PSA is measured by ng/ml PSA levels of 4.0 ng/mL and lower were considered
Measurement of The International Index of Erectile Function (IIEF) in both groups | for each case in both groups the investigator assess IIEF at 6, 12, and 24 months after procedures through study completion, an average of 2 years
  After 6, 12, and 24 months of operation, the questioner is performed. The IIEF-5 score is the sum of the ordinal responses to the 5 items. 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction
Measurement of The Prostate size | for each case in both groups the investigator assess prostate size at 24 months after procedures through study completion, an average of 2 years
  the prostate size was measured by grams by Trans-rectal ultra sound
The operative time of both groups | for each case in both groups the investigator assess the time of operation from induction of anaesthesiatill the end of the operation through study completion, an average of 2 years
  the operative time was measured by minutes in both groups.
Post operative hospital stay time in both groups | for each case in both groups the investigator assess the hospital time from the day of admission of the patient in hospital to do intervention till discharge from hospital through study completion, an average of 2 years
  the Post operative hospital stay time was measured by hours in both groups.
Incidence of The catheter duration post operative in both groups | for each case in both groups the investigator assess the catheter duration from the end of the operation till removal through study completion, an average of 2 years
  The catheter duration was measured by days in both groups.
Measurement of Post operative residual urine (PVR) | for each case in both groups the investigator assess prostate size at 6, 12 and 24 months after procedures through study completion, an average of 2 years
  PVR was measured by ml by pelvi abdominal ultra sound in both groups. Normal ranges are below 150 ml of urine.

SECONDARY OUTCOMES:
Incidence of complications | through two years
  For each case in both groups the investigator assess the safety using incidence of complications by The Clavien-Dindo system

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sa salem, MD, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixon CM, Cedano ER, Pacik D, Vit V, Varga G, Wagrell L, Larson TR, Mynderse LA. Two-year results after convective radiofrequency water vapor thermal therapy of symptomatic benign prostatic hyperplasia. Res Rep Urol. 2016 Nov 21;8:207-216. doi: 10.2147/RRU.S119596. eCollection 2016. PMID 27921028
- [Background] Elshal AM, Soltan M, El-Tabey NA, Laymon M, Nabeeh A. Randomised trial of bipolar resection vs holmium laser enucleation vs Greenlight laser vapo-enucleation of the prostate for treatment of large benign prostate obstruction: 3-years outcomes. BJU Int. 2020 Dec;126(6):731-738. doi: 10.1111/bju.15161. Epub 2020 Sep 30. PMID 32633020
- [Background] Samir M, Tawfick A, Mahmoud MA, Elawady H, Abuelnaga M, Shabayek M, Youssef AEH, Tawfeek AM. Two-year Follow-up in Bipolar Transurethral Enucleation and Resection of the Prostate in Comparison with Bipolar Transurethral Resection of the Prostate in Treatment of Large Prostates. Randomized Controlled Trial. Urology. 2019 Nov;133:192-198. doi: 10.1016/j.urology.2019.07.029. Epub 2019 Aug 9. PMID 31404581
- [Background] McVary KT, Rogers T, Roehrborn CG. Rezum Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology. 2019 Apr;126:171-179. doi: 10.1016/j.urology.2018.12.041. Epub 2019 Jan 21. PMID 30677455
- [Background] Parsons JK, Dahm P, Kohler TS, Lerner LB, Wilt TJ. Surgical Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA Guideline Amendment 2020. J Urol. 2020 Oct;204(4):799-804. doi: 10.1097/JU.0000000000001298. Epub 2020 Jul 23. PMID 32698710
- [Background] Nickel JC, Aaron L, Barkin J, Elterman D, Nachabe M, Zorn KC. Canadian Urological Association guideline on male lower urinary tract symptoms/benign prostatic hyperplasia (MLUTS/BPH): 2018 update. Can Urol Assoc J. 2018 Oct;12(10):303-312. doi: 10.5489/cuaj.5616. No abstract available. PMID 30332601
- [Background] Bole R, Gopalakrishna A, Kuang R, Alamiri J, Yang DY, Helo S, Ziegelmann MJ, Kohler TS. Comparative Postoperative Outcomes of Rezum Prostate Ablation in Patients with Large Versus Small Glands. J Endourol. 2020 Jul;34(7):778-781. doi: 10.1089/end.2020.0177. Epub 2020 Jun 12. PMID 32408768
- [Background] Garden EB, Shukla D, Ravivarapu KT, Kaplan SA, Reddy AK, Small AC, Palese MA. Rezum therapy for patients with large prostates (>/= 80 g): initial clinical experience and postoperative outcomes. World J Urol. 2021 Aug;39(8):3041-3048. doi: 10.1007/s00345-020-03548-7. Epub 2021 Jan 3. PMID 33392646
- [Background] Elterman D, Bhojani N, Vannabouathong C, Chughtai B, Zorn KC. Rezum therapy for >/=80-mL benign prostatic enlargement: a large, multicentre cohort study. BJU Int. 2022 Oct;130(4):522-527. doi: 10.1111/bju.15753. Epub 2022 May 7. PMID 35466513